CLINICAL TRIAL: NCT02125019
Title: Longitudinal Evaluation of Taxane Induced Neuropathy in Early Stage Breast Cancer
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Nicole Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-13010
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Taxane; Gait; Men; Women
MeSH Terms: conditions — Breast Neoplasms; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients: This is a single arm study evaluating feasibility of evaluating gait and parameter changes in patients with early stage breast cancer undergoing adjuvant taxane chemotherapy.

SUMMARY:
Longitudinal Evaluation of Taxane induced neuropathy in early stage breast cancer.

DETAILED DESCRIPTION:
A study assessing the feasibility of evaluating neuropathy symptoms prospectively using testing of gate and balance parameters.

ELIGIBILITY:
Inclusion criteria

* Patients (men and women) diagnosed with breast cancer stages I-III initiating first line adjuvant or neoadjuvant therapy with paclitaxel or docetaxel
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with functional limitations due to musculoskeletal conditions can be included, because these conditions are known to remain stable over the relatively short duration of the study.
* Concurrent standard and investigational agents are permissible with the standard chemotherapy drugs.

Exclusion Criteria

* Prior known chemotherapy or targeted therapy (for breast cancer or other malignancies that is known to be associated with neuropathy in the last 12 months(platinum therapy, bortezomib, vinblastine, etc.)
* Prior taxane exposure at any time
* Preexisting known diagnosis of any type of neuropathy prior to start of paclitaxel or docetaxel chemotherapy
* Pregnant or nursing women.
* Unable to give informed consent.
* Preexisting lower extremity amputation
* Inability to walk or stand without assistance due to any condition
* Neuropathic pain medications prior to start of study including gabapentin, pregabalin, amytriptyline, and duloxetine (but initiation of neuropathic pain medications during treatment are permissible)
* Patients needing ambulatory assist devices
* Back or lower extremity surgery in the last 6 months
* Back or lower extremity surgery at any timepoint that interferes with gait and balance per patient or provider report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with breast cancer stages I-III
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Identify gait and balance parameters that are affected by during adjuvant/neoadjuvant taxane (paclitaxel or docetaxel) chemotherapy. | Up to 2 years

SECONDARY OUTCOMES:
Evaluate the natural history of changes in these gait and balance parameters and their relationships with validated self-reported assessment tools of CIPN such as CIPN-20 and TNS | Up to 2 years
Identify gait and balance changes as a consequence of chemotherapy with paclitaxel or docetaxel in the laboratory measuring the motion of the entire body in three dimensions with great accuracy. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Williams, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu